CLINICAL TRIAL: NCT05102760
Title: Pericapsular Nerve Group (PENG) Block vs. the Fascia Iliaca Compartment (FIC) Block for Patients With Isolated Hip Fractures in the Emergency Department
Brief Title: PENG vs. FIC Block for Hip Fracture ED Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-02-09
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pain; Hip Fracture
Keywords: Pain; Hip Fracture; Nerve Block; Ultrasound
MeSH Terms: conditions — Pain; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia Iliaca Compartment (Active Comparator): Fascial Iliaca block (FIC) (40mL of Bupivacaine 0.25%) for patients with hip fractures in the ED
  Interventions: Procedure: Nerve Block using FIC Proceedure
- PENG Block (Active Comparator): Pericapsular Nerve Group (PENG) Block (20mL of Bupivacaine 0.50%)
  Interventions: Procedure: Nerve Block using PENG Proceedure

INTERVENTIONS:
Procedure: Nerve Block using FIC Proceedure — Ultrasound Guided Nerve Block for Hip Fracture Patients using the FIC Proceedure
  Arms: Fascia Iliaca Compartment
Procedure: Nerve Block using PENG Proceedure — Ultrasound Guided Nerve Block for Hip Fractures Patients using the PENG Procedure
  Arms: PENG Block

SUMMARY:
Ultrasound-guided nerve blocks are an important tool for treating pain due to orthopedic injury in the ED. They provide long lasting, opioid-sparing pain relief that is generally safe and well-tolerated by patients1. Elderly patients with hip fractures commonly present to the ED, and their injury can be painful. Commonly used opioid pain regimens can have deleterious side effects, especially in elderly patients, like somnolence, delirium, hypotension and respiratory depression.

The fascia iliaca compartment (FIC) block has become a familiar technique to emergency physicians as a pain control treatment for hip fractures. The pericapsular nerve group (PENG) block has recently been proposed as a novel method to treat pain due to hip, acetabular and pelvic fracture by targeting the terminal sensory articular nerve branches of the femoral nerve (FN), obturator nerve (ON), and accessory obturator nerve (AON). At this time there has been no study comparing the efficacy of the two nerve blocks, PENG and FIC.

This aim of this study is to compare the efficacy of the PENG block (20mL of Bupivacaine 0.50%) to that of the FIC block (40mL of Bupivacaine 0.25%) for patients with hip fractures in the ED. Our hypothesis is that PENG will demonstrate analgesia that is non-inferior to FIC. Subjective pain scores on a scale of 0 to 10 will be assessed before and after the block. All subjects will receive 4mg of morphine after consent and prior to the block.

DETAILED DESCRIPTION:
Ultrasound-guided nerve blocks are an important tool for treating pain due to orthopedic injury in the ED. They provide long lasting, opioid-sparing pain relief that is generally safe and well-tolerated by patients1. Elderly patients with hip fractures commonly present to the ED, and their injury can be painful. Commonly used opioid pain regimens can have deleterious side effects, especially in elderly patients, like somnolence, delirium, hypotension and respiratory depression.

The fascia iliaca compartment (FIC) block has become a familiar technique to emergency physicians as a pain control treatment for hip fractures. The pericapsular nerve group (PENG) block has recently been proposed as a novel method to treat pain due to hip, acetabular and pelvic fracture by targeting the terminal sensory articular nerve branches of the femoral nerve (FN), obturator nerve (ON), and accessory obturator nerve (AON). At this time there has been no study comparing the efficacy of the two nerve blocks, PENG and FIC.

This aim of this study is to compare the efficacy of the PENG block (20mL of Bupivacaine 0.50%) to that of the FIC block (40mL of Bupivacaine 0.25%) for patients with hip fractures in the ED. Our hypothesis is that PENG will demonstrate analgesia that is non-inferior to FIC. Subjective pain scores on a scale of 0 to 10 will be assessed before and after the block. All subjects will receive 4mg of morphine after consent and prior to the block.

A secondary aim is to show that the PENG block is preferable to the FIC block because it does not target motor nerves, thus preserving motor function allowing for an accurate neurological exam and hopefully providing for earlier ambulation. Also, we aim to determine if PENG block results in an significant reduction in amount of systemic pain medication needed for the patient.

This is a single-centered, prospective, randomized, blinded study involving patients who present to the ED with an isolated hip fracture. Patients who meet inclusion criteria will be consented for the study and then randomized to receive either a FIC block or a PENG block. Patients who are potentially to be enrolled in the study will receive standardized systemic analgesia while awaiting x-rays. If needed, patients will be administered morphine for breakthrough pain after the nerve blocks are placed. The exception to this standardization will be patients with a morphine allergy.

The research associate will screen for patients and confirm with the attending physician that the subject is eligible for enrollment and is able to give consent. The patient consented by a member of the research team, who will assess the patient's pain score on a scale of 0 to 10 prior to the block. The patient will then be randomized to receive either the FIC block or the PENG block to be performed by a member of the ultrasound faculty. The research associate will be blinded to the type of block being performed by the ultrasound faculty member. The research associate will then reassess the patient's pain score on the 0-10 scale at the 30 minute and 60-minute mark. They will also assess for any adverse events after the block is performed. The research associate will note the motor function in the quadriceps muscle 30 min and 60 min after the nerve block is placed. Any rescue medication given after the nerve block is placed in the ED will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult Emergency Medicine Patients over 18 years of age
* Isolated hip fracture, intertrocanteric or more proximal
* Pain score 5 or greater on a scale of 0 to 10 just prior to nerve block placement

Exclusion Criteria:

* Patients with multi-system trauma
* People who are unable to communicate their level of pain\
* Pregnant patients
* Pediatric Patients (less than 18 years of age)
* Intoxicated Patients
* Abnormal Vital Signs (HR>120bpm, MAP <65, Pulse Ox <95%)
* Patients on long term systemic opioid analgesia
* Allergy to amide local anesthetics

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Score at 30 Minutes | 30 minutes post administration of nerve block
  The pain score at 11 point Likert Scale ranging 0 (no pain) to 10 (very severe pain) at 30 minutes post nerve block procedure

SECONDARY OUTCOMES:
Pain Score at 60 minutes | 60 minutes post administration of nerve block
  The pain score at 11 point Likert Scale ranging 0 (no pain) to 10 (very severe pain) at 60 minutes post nerve block procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Haines, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT05102760/Prot_SAP_000.pdf